CLINICAL TRIAL: NCT04981418
Title: Evaluating the Management of Chronic Pelvic Girdle Pain Following Pregnancy (EMaPP): A Randomised Controlled Feasibility Trial
Brief Title: Evaluating the Management of Chronic Pelvic Girdle Pain
Acronym: EMaPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: Royal Cornwall Hospitals Trust (Other); University Hospital Plymouth NHS Trust (Other)
Responsible Party: Principal Investigator, Bradley Halliday, Teaching and research associate, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 297938
Record Dates: First submitted 2021-07-01; First posted 2021-07-29 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Orthotic Devices; Exercise; Counseling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All outcomes measures are collected via self report means. This will enable the investigators to be blinded to the outcomes measures reported. Treating clinicians are also blinded to the outcome assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): will receive standardised advice on management of pelvic girdle pain, through a discussion centred around 'Guidance for Mothers-to-be and New Mothers: Pregnancy-related Pelvic Girdle Pain' booklet (https://pogp.csp.org.uk/system/files/pogp-pgppat_3.pdf). This publicly available, specialist physiotherapy approved, standardised leaflet, provides information reflective of current best practice. The participant can use this as an ongoing resource. The physiotherapist will teach participants a standardised programme of exercises, typical of those provided within usual physiotherapy practice. Written explanation/illustrations of these exercises will be provided and the women asked to undertake these at home, three times/week.
  Interventions: Other: Exercise; Other: advice
- Intervention group (Experimental): In addition to the control groups intervention of exercise and advice, women in the intervention group will be fitted with the customised pelvic support shorts (DM Orthotics Ltd, https://www.dmorthotics.com).
  Prior to the first physiotherapy session, those women allocated to the intervention group will have recieved the support shorts in the post together with standardised written information on wear time/washing. At the first physiotherapy session (one hour), the woman will be asked to try them on so that the physiotherapist can review the fit and comfort of the shorts. The physiotherapist will reinforce the written advice about wear time and care of the shorts, and answer any queries / brainstorm any issues. At session two (30 minutes), ~10 days later, the physiotherapist will review the fit and wearing of the shorts, problem solve any issues that have arisen, and review exercises to ensure they are being performed correctly.
  Interventions: Device: customised pelvic support shorts; Other: Exercise; Other: advice

INTERVENTIONS:
Device: customised pelvic support shorts — These apply targeted compressive forces to the pelvic girdle through selective precisely positioned reinforced lycra panels that aim to stabilize and align body segments to improve function and reduce unwanted movements. The construction material (Nylon and Elastane) is durable and breathable, and its mechanical properties enable it to provide "dynamic" stability and support (rather than the rigid support provided by "off-the-shelf" belts) during movement/functional activities. This aims to optimise comfort and movement to increase wear compliance, which is crucial as any benefits gained rely upon this.
  Other Names: DEFO; ORTHOTIC
  Arms: Intervention group
Other: Exercise — Women will be provided with up to a maximum of 4 exercises from a pre-defined list of exercises. Suggested dosages are referred to in the protocol. The exercise programme contains a range of exercise focused around the pelvic girdle and hips (including movement control and strengthening
Other: advice — standardised advice on management of pelvic girdle pain, through a discussion centred around 'Guidance for Mothers-to-be and New Mothers: Pregnancy-related Pelvic Girdle Pain' booklet (https://pogp.csp.org.uk/system/files/pogp-pgppat_3.pdf). This publicly available, specialist physiotherapy approved, standardised leaflet, provides information reflective of current best practice. The participant can use this as an ongoing resource.

SUMMARY:
Evaluating the Management of chronic Pelvic girdle pain following Pregnancy (EMaPP)

During pregnancy pelvic girdle pain is common. This pain will often reduce following childbirth, however almost 20% of women continue to suffer significant pain for at least three months afterwards. When pain is severe it will affect everyday activities and quality of life. Usual treatment typically involves Physiotherapy (advice and exercise) and provision of an "off the shelf" rigid pelvic support belt. Women often find these uncomfortable and difficult to use. A customised pelvic orthotic (referred to as pelvic support shorts) is an alternative that on initial testing has shown promising results in women with chronic pelvic girdle pain.This feasibility study aims to obtain the data and operational experience necessary to inform the conduct and finalise the design of a future large randomised controlled trial. The investigators will also gather women's views about the support shorts and the trial. It is vital to understand what treatments are beneficial to this group of women and this is the main driver for this National Institute of Health Research funded trial.

Following screening and consent, 60 women aged > 18 years, with severe, persistent post-partum pelvic girdle pain will be recruited into the trial. They will be randomised to receive either usual care (advice and exercise) or usual care and the customised pelvic support shorts. All women will receive 2 web-based sessions with a physiotherapist who will provide this intervention. All will complete web-based self-report questionnaires (pain, function, quality of life, continence, depression) at baseline, 3 and 6 months. Fortnightly scoring of pain and medication usage throughout the trial timeline complements this. Fifteen women and five clinicians will be interviewed at the end of the trial to explore their experiences of wearing/providing the "support shorts" and participating in the trial.

DETAILED DESCRIPTION:
The investigators will undertake a multi-centre feasibility RCT, randomising participants to receive either the "pelvic support shorts" plus standardised information and exercises (intervention) or standardised information and exercises alone (control).

The investigators will recruit 60 women from the South West of England who are experiencing chronic (≥3 months) and severe pelvic girdle pain following pregnancy.

Following screening and consent, baseline assessment will be undertaken using a range of patient-reported measures: pain, depression, continence, function, quality of life, health/social care and patient resource use. Women will randomly allocated to intervention or control. Two weeks following randomisation, all participants will attend a physiotherapy session via web-conference to receive standardised information and suggested exercises. In addition, intervention group participants will receive two pairs of the pelvic support shorts. In line with usual physiotherapy practice, all participants will receive a follow-up review session via web-conference, approximately 10 days later.

Throughout the study timeframe, medication usage and pain rating scale scores will be completed by the women, on a fortnightly basis, via web-based self-report questionnaires. Additionally, at 12 and 24 weeks all baseline patientreported measures will again be collected. A qualitative sub- study, involving interviews (telephone or web-based) will explore participant experiences of wearing (patient) and providing (physiotherapists) the support shorts, and of the study itself.

The Population

The investigators shall recruit women, 18 and over, experiencing chronic and severe pelvic girdle pain. This pain must have started or been aggravated during pregnancy and have continued for at least three-months following childbirth. The pain is 'severe' if it causes walking or stair climbing to be bothersome and scores positively on a range of pain provocation tests. Potential participants will be excluded if they have pathologies which cause pelvic girdle pain (e.g. infection, trauma), are currently pregnant, report an allergy to Lycra, or where pain has persisted for > two years following pregnancy so that the investigators can limit the risk of other pathologies being the origin of pain.

Intervention and Control.

All treatment will be provided by NHS physiotherapists at two web-based sessions.

Control Group.

Both groups will receive standardised advice on management of pelvic girdle pain, through a discussion centred around 'Guidance for Mothers-to-be and New Mothers: Pregnancy-related Pelvic Girdle Pain' booklet (https://pogp.csp.org.uk/system/files/pogp-pgppat_3.pdf). This publicly available, specialist physiotherapy approved, standardised leaflet, provides information reflective of current best practice. The participant can use this as an ongoing resource. The physiotherapist will teach participants a standardised programme of exercises, typical of those provided within usual physiotherapy practice. Written explanation/illustrations of these exercises will be provided and the women asked to undertake these at home, three times/week.

Intervention Group

In addition to the above, women in the intervention group will be fitted with the customised pelvic support shorts (DM Orthotics Ltd, https://www.dmorthotics.com).

Prior to the first physiotherapy session, those women allocated to the intervention group will have recieved the support shorts in the post together with standardised written information on wear time/washing. At the first physiotherapy session (one hour), the woman will be asked to try them on so that the physiotherapist can review the fit and comfort of the shorts. The physiotherapist will reinforce the written advice about wear time and care of the shorts, and answer any queries / brainstorm any issues. At session two (30 minutes), ~10 days later, the physiotherapist will review the fit and wearing of the shorts, problem solve any issues that have arisen, and review exercises to ensure they are being performed correctly.

After these two appointments all participants will be continue to self-manage the condition for the remainder of the trial. Participants are not prevented from accessing further healthcare. The trial is capturing this information through a resource use questionnaire which is collected at baseline, 12 and 24 weeks.

Outcomes and their measurement.

In our feasibility trial, participants will be requested to complete a range of self-report outcome measures via a mobile/web app. Our PPI discussions led us to choose self-report questionnaires, completed via a web-based application, to minimise burden (time and travel) on our participants who are experiencing significant pain. This is particularly important since driving and travelling frequently exacerbated this pain. Some women may prefer paper versions, returned by post.

In line with the remit of a feasibility trial, the investigators include a variety of measures to determine their performance in the context of this trial and, along with trial participants and our PPI group, to identify those that may be most appropriate for the definitive trial. All are standardised patient-report measures which have been previously used in studies investigating pelvic girdle pain.

Demographic data will be collected at screening (age, weight, number of pregnancies, severity/duration/site of pain).

Additional clinical data will be collected at baseline: medication, week of delivery, length of labour, induction required, mode of delivery, episiotomy/perineal tear, baby's gender and weight, presence/absence of back pain prior to pregnancy.

All outcome measures will be completed at baseline and 12 and 24 weeks following the first intervention session, apart from the Pain Rating Scale and medication usage which will be completed fortnightly.

Recruitment Procedure

Women will be recruited from three NHS Trusts across the Southwest of England:

1. Royal Cornwall NHS Foundation Trust, Cornwall Partnership NHS Foundation Trust, and University Hospitals Plymouth NHS Trust. Physiotherapists in musculoskeletal outpatient and women's health services will be key recruiters due to their contact with women experiencing chronic pain following pregnancy. They will raise study awareness and provide patients with study information leaflets. The Clinical Research Network (CRN) staff will undertake a database search, eligibility check, and mail-out to potential participants. With the clients' consent, the CRN nurse will inform the research team of potential participants via a study specific email account. The research team will telephone/email the potential participant to undertake initial screening and, if still apparently eligible, book a web-based screening appointment.
2. Research active general practices with an on-site First Contact Physiotherapy Practitioner. CRN staff will undertake a database search and mail-out to potentially eligible patients, inviting them to express an interest in the trial. With the consent of those interested, names will be forwarded to the research team.

The study will be advertised in local children's centres and on social media [Mumsnet; facebook pages of the Pelvic Partnership Pelvic Girdle Pain Support Group, National Maternity Voices, National Childbirth Trusts], and via relevant hospital web-site and twitter accounts which advertise research trials.

A research physiotherapist will undertake the web-based screening/measurement for shorts and baseline assessments, in separate sessions independent of treatment. The nature of the self-report measures ensures the assessor will not influence participant responses. Participants will be asked not to discuss their treatment with the researcher.

Randomisation and blinding.

Following baseline assessment, the research physiotherapist will enter key participant details (number of pregnancies, pain onset/duration) into the Clinical Trial Unit's (CTU) web-based randomisation system and immediately receive that participant's group allocation. Randomisation will be stratified by centre and presence/absence of back pain pre- pregnancy. An automatic email will be sent by the CTU to the NHS-treating physiotherapist to inform them of the woman's group allocation, and enable them to schedule an outpatient appointment approximately two weeks (+/-1 week) later. A second email with the patient's measurements will be sent to DM Orthotics Ltd to allow manufacture of the customised shorts.

Sample size

The investigators aim to recruit 60 participants over 7-months. As this proposal is for a feasibility trial, a sample size calculation is not appropriate. Instead, the investigators aim to sample sufficient participants to provide the operational experience to conduct a larger trial and to provide data to inform future sample size calculation.

EMBEDDED QUALITATIVE COMPONENT.

Qualitative research to explore "real-life" experience is important in order to understand and learn from participants about whether trial processes, the intervention and outcome measures are acceptable. The investigators will therefore undertake interviews with a sub-sample of women to explore the:

* acceptability of trial methods across both trial arms
* acceptability (comfort, wear-time) of the support shorts
* impact the intervention may/may not have on women's lives.
* adherence to the exercise regime over the course of the trial

Ten purposively sampled participants from the trial will include 5 trial participants randomised to the control group and 5 participants from the intervention group. These will include women receiving interventions from both the secondary care (RCHT & UHP) and primary care sites (GP practices). This will be run through individual one off semi-structured telephone interviews using a topic guide. Interviews will occur at the end of the trail period.

Five NHS physiotherapists (from secondary and primary care sites) involved within the trial will be purposively sampled to provide information on the acceptability of the trial methods across both trial arms.

ECONOMIC EVALUATION. The investigators will estimate the resource requirements of the intervention, and establish the framework for a future cost effectiveness analysis alongside a full RCT. Data on intervention resources will be collected about participant-level contact and non-contact time, and training for delivery staff. Participants will self-report health, social and wider care resource use, using the Resource Use Questionnaire from our antenatal study and adapted for this trial by our PPI Group.

ELIGIBILITY:
Inclusion Criteria:

* Women aged greater than or equal to 18
* Able and willing to provide informed consent
* Self reported Persistent pelvic girdle pain (PGP) (≥3 months post partum)
* Self reported severe PGP (causing walking or stair climbing to be bothersome)
* Diagnosed with PGP in line with European guidelines
* PGP must have started or been aggravated during pregnancy, as determined by self report

Exclusion Criteria:

* known allergy to lycra
* age < 18
* currently pregnant
* PGP for > 2 years post partum
* Self reported history of pathologies causative of lumbo pelvic pain(e.g. Infection, trauma, cancer)
* Participating in concurrent interventional research which may over-burden the patient or confound data collection
* There are no special arrangements made for participants who are unable to adequately understand verbal and/or written English. There is no intention to exclude patients, therefore, if they have regular access to a friend or family member who is able to translate for them they would be able to participate
* Participants who lack capacity to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women only. This study is investigating pregnancy related pelvic girdle pain. The participants will need to have self reported PGP and therefore be female.
Enrollment: 24 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-02-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline pain intensity (Numerical Rating Pain Scale) at 24 weeks | up to 24 weeks
  Numerical pain rating scale. This is to assess pain levels across the course of the study period of 24 weeks.
  Women will be asked to rate their pain experience over the past fortnight, using the NPRS, in four categories:
  * Worst level of pelvic pain during the day
  * Average level of pelvic pain during the day
  * Worst level of pelvic pain during the night
  * Average level of pelvic pain during the night
  Scale runs between 0-10. Higher scores represent greater pain intensity.

SECONDARY OUTCOMES:
Pelvic girdle questionnaire | Baseline, 12 weeks, 24 weeks
  The PGQ is a condition-specific instrument that assesses activity limita-tions (PGQ activity with 20 items) and symptoms (PGQ symptom with 5 items) in women with PGP during pregnancy as well as postpartum. Items are scored on a 4-point descriptive scale (0-3).
  All scores are summarized and divided by the to-tal possible score of 75 (maximum pos-sible scores of 60 for activity and 15 for symptoms), subsequently recalculated to a percentage, resulting in percentage scores ranging from 0 (no disability) to 100 (severe disability).
EQ-5D-5L | Baseline, 12 weeks, 24 weeks
  Evaluation of Quality of life
SF36 | Baseline, 12 weeks, 24 weeks
  Short form 36 Evaluation of Quality of life
EPDS | Baseline, 12 weeks, 24 weeks
  Edinburgh Post Natal Depression Scale This is the most commonly used, validated self-report screening tool for post-natal depression. Comprising 10 questions rating feelings over the past 7-days, it is easy to complete, with good diagnostic accuracy at a cut-off of ≥11 points.
  Higher scores represent more likely depression.
iciq-ui sf | Baseline, 12 weeks, 24 weeks
  International Consultation on Incontinence Questionnaire - Urinary incontinence - Short Form,
  It comprises questions regarding frequency/amount of urine leakage, and interference with everyday life. It obtains a brief yet comprehensive summary of the level, impact and perceived cause of the symptoms of incontinence.
Support shorts wear time | 24 weeks
  For the intervention group wear-time will be determined by a sensor sewn into the seam of the support shorts (able to distinguish wear-time from washing/drying cycles , Orthotimer Ltd, www.orthotimer.com). After the 6-month trial, women will be asked to remove the sensor and post it back to the research team (FREEPOST envelope) for them to download the data and analyse it.
Health resource use questionnaire | Baseline, 12 weeks, 24 weeks
  Data on health, social and wider care resource use will be collected using a self-report resource use questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Freeman, PhD, Principal Investigator — University of Plymouth
Locations (1):
- University Hospitals Plymouth NHS Trust, Derriford Hospital, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to the final trial dataset
  Data generated as a result of this trial will be available for inspection on request by the EMaPP research team, University of Plymouth representatives, the REC, local R&D Departments and regulatory authorities
Supporting Information: Study Protocol, CSR
Time Frame: Academic paper to be written on completion of trial. Expected completion May 2022